CLINICAL TRIAL: NCT01282736
Title: Comparison of Integrative Response Therapy and Cognitive Behavioral Therapy Guided Self-Help for Binge Eating Disorder
Brief Title: Guided Self-Help for Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SU-01122011-7362
Record Dates: First submitted 2011-01-14; First posted 2011-01-25 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Binge Eating Disorder
Keywords: eating disorder; binge eating
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders; Bulimia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrative Response Therapy (Experimental): IRT is based on affect regulation theories of binge eating and adds emphasis on cognitive restructuring techniques. IRT is a 10 session, group-based, guided-self-help treatment that works to decrease binge eating by primarily enhancing emotion coping skills, in addition to transforming faulty interpretations and reducing vulnerabilities (e.g., interpersonal events) that risk overwhelming emotion and problematic cognitions.
  Interventions: Behavioral: Integrative Response Therapy
- Cognitive Behavioral Therapy (Active Comparator): Cognitive Behavioral Therapy guided self-help (CBT-GSH), based on the restraint model of binge eating, has been adapted from individual format to a 10 session, group-based therapy for the purpose of this study. The book 'Overcoming Binge Eating' is employed in the present study and consists of Part 1, an educational background on BED, and Part 2, a 6 step treatment program to overcome binge eating.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Integrative Response Therapy — A 10 session manualized version of IRT is employed . Each of the 10 group therapy sessions will be 60 minutes in length. Non-specialty trained Masters-level therapists will lead IRT after undergoing IRT training with the PI.
  Arms: Integrative Response Therapy
Behavioral: Cognitive Behavioral Therapy — A 10 session manualized version of CBT-GSH is employed . Each of the 10 group therapy sessions will be 60 minutes in length. Non-specialty trained Masters-level therapists will lead CBT-GSH after undergoing CBT-GSH training with the PI.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The proposed study will employ a randomized design to evaluate the efficacy of two group-based guided self-help treatments: Integrative Response Therapy (IRT) and Cognitive Behavior Therapy Guided Self-Help, a treatment of known efficacy, in group-format (CBT-GSHg) in the treatment of Binge Eating Disorder (BED), and explore (1) moderators and mediators of treatment, (2) the relative cost-effectiveness of the two treatments, and (3) between group differences on secondary measures (e.g., eating disorder and general psychopathology).

DETAILED DESCRIPTION:
The focus of this proposal is on BED among an adult population. Guided self-help treatments (GSH) for BED appear promising and may be more readily disseminated than efficacious specialty treatments such as Cognitive Behavioral Therapy (CBT) and Interpersonal Psychotherapy (IPT) given the latter's administration costs and time requirements. The proposed study uses a new group-based, guided self-help BED treatment called Integrative Response Therapy (IRT). IRT is primarily based upon the affect regulation theory of binge eating (e.g., binge eating is an attempt to alter distressing emotional states), while adding cognitive restructuring techniques. IRT teaches effective ways to cope with aversive emotions and reframe faulty cognitions while reducing vulnerabilities that are likely to lead to problematic emotional responding & cognitions such as physical needs (e.g., hunger, sleep deprivation), interpersonal conflict, and, when possible, unpleasant external events. IRT's primary goal is to significantly decrease episodes of binge eating and associated eating disorder pathology.

CBT-GSH is a frequently used manual-based form of GSH that has demonstrated efficacy. CBT, based on the restraint model, intervenes via behavioral techniques to replace restrained eating with more regular eating patterns and cognitive techniques to restructure an individual's problematic thoughts that over-evaluate shape and weight. Research literature indicates that CBT-GSH is a viable self-help BED treatment that appears to be superior to wait-list control conditions, equivalent to IPT, a specialty treatment, and superior to Behavioral Weight Loss treatment at 2-year follow-up. There are then, a number of reasons for further research on GSH in general and CBT-gsh specifically.

The proposed study will lay the groundwork for identifying which GSH treatment should be investigated in a subsequent, larger trial that would evaluate a clinically relevant algorithm for the treatment of BED.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV research criteria for Binge Eating Disorder (although frequency criteria will be lessened to that proposed in DSM-V;1 time per week for 3 months).
* Be male or female between 18 and 75 years.
* Be available and committed to attend full treatment and follow-up
* Adequate transportation to the clinic.
* Be literate in English (this is required for inclusion because sessions will be conducted in English and written and visual materials are in English).
* Have a Primary Health Care Provider.

Exclusion Criteria:

* Current psychosis or severe depression with suicidal risk; a severity that would likely require additional psychotherapeutic or psychopharmacologic treatment or interfere with participation in this group therapy or with day to day functioning. Depressive disorders not meeting the intensity factor of the exclusion criteria may be entered to the study.
* Current Anorexia or Bulimia Nervosa or purging behaviors over the past six months.
* Current drug and/or alcohol abuse/dependence.
* Current medication primarily indicated for its effect on appetite or weight, unless the participant is willing to withdraw from such medications under supervision of their primary care physician.
* Current chemotherapy.
* Current participation in psychotherapy, unless the participant is willing to discontinue treatment.
* Psychotropic medication use, including antidepressants, are acceptable if doses were stable for at least 1 month prior to assessment.
* Pregnant or plans to become pregnant within the next 12 months.
* BMI greater than 45.
* Planning to have Bariatric surgery within the next 12 months.
* No transportation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
number of binge days over the previous 28 days | 16 weeks post-treatment
  Assessed via the Eating Disorder Examination

SECONDARY OUTCOMES:
emotion driven urges to eat | 16 weeks post-treatment, 6 and 12 month follow-up
  Assessed via the Emotional Eating Scale
adaptation time intervals and response accuracy for emotion related stimuli | 16 weeks post-treatment
  Assessed via the Emotion Conflict Adaptation Task
depression | 16 weeks post-treatment, 6 and 12 month follow-up
  Assessed via the Beck Depression Inventory
self-esteem | 16 weeks post-treatment, 6 and 12 month follow-up
  Assessed via the Rosenberg Self-Esteem Scale
quality of life | post-treatment, 6 and 12 month follow-up
  Assessed via the Quality of Well-Being Scale
use of health services | at (approximately) 1 month intervals throughout 16 week intervention (4 times total)
  Assessed via the Health Care Diary

CONTACTS AND LOCATIONS:
Overall Officials: Athena Robinson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States